CLINICAL TRIAL: NCT01285648
Title: APPLICATION OF CONTINUOUS POSITIVE AIRWAY PRESSURE IN POSTOPERATIVE OF LUNG RESECTION
Brief Title: Study of CPAP as Intervention After Lung Resection
Acronym: CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: APPLICATION OF CONTINUOUS POSITIVE AIRWAY PRESSURE IN POSTOPERATIVE OF LUNG RESECTION, Unicamp
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ROCETO130682
Record Dates: First submitted 2011-01-25; First posted 2011-01-28 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Lung Cancer; Pulmonary Complications
Keywords: chest tubes,; Continuous Positive Airway Pressure,; lung resection, thoracic surgery,; noninvasive ventilation,; postoperative
MeSH Terms: conditions — Lung Neoplasms | interventions — Continuous Positive Airway Pressure; Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cpap (Other): This group joined chest physiotherapy with CPAP via nasal masks for two hours.CPAP was continued from the immediate postoperative day until the second postoperative day, twice a day.
  Interventions: Procedure: Cpap
- Chest Physiotherapy (Other): Chest Physiotherapy consisted of bronchial hygiene techniques and pulmonary expansion, in addition to exercises, and received oxygen supplementation to maintain the pulse oxymetry saturations > 90%.
  Interventions: Procedure: Cpap

INTERVENTIONS:
Procedure: Cpap — This study did not involved drugs. The Oxygenation index, Borg Scale, pain scale and the presence and duration of thoracic drainage was determined in the immediate postoperative (POi) period and in the first and second postoperative (PO1, PO2) days in 40 patients who underwent elective lung resection,in two groups of intervention: chest physiotherapy, and associate this with cpap
  Other Names: Noninvasive ventilation; lung resection

SUMMARY:
The aim of this study was to compare the oxygenation index (OI), dyspnea, and pain scale and evaluate the duration of thoracic drainage and pleural air leaks after lung resection in two groups of patients: chest physiotherapy (CP) patients and combined CP and Continuous Positive Airway Pressure (CPAP) patients.

DETAILED DESCRIPTION:
In pulmonary resection surgery complications that lead to significant functional losses of the lung parenchyma and alterations in the ventilatory function may trigger retention of secretions, atelectasis, pneumonia and respiratory failure, which prolong the duration of mechanical ventilation and hospitalisation and contribute to the increase in risk of mortality.

In this study the oxygenation index (OI), Borg Scale, pain scale and the presence and duration of thoracic drainage was determined in the immediate postoperative (POi) period and in the first and second postoperative (PO1, PO2) days in 40 patients who underwent elective lung resection.

Similar to Chest Physiotherapy, the preventive application of CPAP in the postoperative period after lung resection in our study also appeared to be a safe technique, which allowed improved oxygenation without increasing air leaks through the thoracic drains.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of lung cancer and an indication for lung resection (lobectomy, bilobectomy and pneumonectomy) with posterolateral thoracotomy;
* aged between 40 and 75 years.

Exclusion Criteria:

* Patients who refused to participate in the survey;
* lung resection with incisions other than posterolateral;
* patients who had contraindications to the use of noninvasive ventilation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Bubbling drains | From immediate postoperative until fifth, along the study, in a total of one year
  From the immediate postoperative day until hospital discharge, the presence of chest tubes and the occurrence of air leaks in them as evidenced by the bubbling of the water seal were recorded. The maintenance and removal of drains or their use with wall suction were determined by applying the medical protocol of the institution through the analysis of X-rays and the amount of drained fluid.

SECONDARY OUTCOMES:
Pain score | Reported pain score after lung resection, along the study, during one year
  Before beginning the chest physiotherapy protocols, the patient was asked to rate their pain from zero to ten according to its intensity (the larger the score, the greater the intensity of pain).

CONTACTS AND LOCATIONS:
Overall Officials: Lígia S. Roceto, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Campinas State University, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Roceto Ldos S, Galhardo FD, Saad IA, Toro IF. Continuous positive airway pressure (CPAP) after lung resection: a randomized clinical trial. Sao Paulo Med J. 2014;132(1):41-7. doi: 10.1590/1516-3180.2014.1321525. PMID 24474079